CLINICAL TRIAL: NCT03653299
Title: Acute Effects of Phototherapy With Combination of Super-pulsed Laser and LEDs on Gait and Balance of Post-stroke Individuals: A Randomized, Controlled and Triple-blind, Clinical Trial
Brief Title: Effects of Phototherapy on Gait and Balance of Post-stroke Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adriane Aver Vanin, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CEP-211286
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Post-stroke in Association to Phototherapy
Keywords: stroke; phototherapy; gait; balance; functional mobility
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A - Placebo, 10J, 30J and 50J (Experimental): The phototherapy will be divided in programs 1, 2, 3 and 4. One of these programs will consist in placebo and the others in active phototherapy 10J, 30J and 50J.
  The subjects allocated in group Phototherapy A will receive the programs in the following order 1, 2, 3 and 4, before the tests.
  Interventions: Device: Placebo or Active Phototherapy (MR4)
- Group B - Placebo, 10J, 30J and 50J (Experimental): The phototherapy will be divided in programs 1, 2, 3 and 4. One of these programs will consist in placebo and the others in active phototherapy 10J, 30J and 50J.
  The subjects allocated in group Phototherapy B will receive the programs in the following order 2, 3, 4 and 1, before the tests.
  Interventions: Device: Placebo or Active Phototherapy (MR4)
- Group C - Placebo, 10J, 30J and 50J (Experimental): The phototherapy will be divided in programs 1, 2, 3 and 4. One of these programs will consist in placebo and the others in active phototherapy 10J, 30J and 50J.
  The subjects allocated in group Phototherapy C will receive the programs in the following order 3, 4, 1 and 2, before the tests.
  Interventions: Device: Placebo or Active Phototherapy (MR4)
- Group D - Placebo, 10J, 30J and 50J (Experimental): The phototherapy will be divided in programs 1, 2, 3 and 4. One of these programs will consist in placebo and the others in active phototherapy 10J, 30J and 50J.
  The subjects allocated in group Phototherapy D will receive the programs in the following order 4, 1, 2 and 3, before the tests.
  Interventions: Device: Placebo or Active Phototherapy (MR4)

INTERVENTIONS:
Device: Placebo or Active Phototherapy (MR4) — Phototherapy, placebo or active, will applied in 9 different points of anterior muscle of the thigh, 6 different points of posterior muscle of the thigh and 2 different points of the gastrocnemius muscle, bilaterally. Once a week during for 4 weeks, before the tests, the phototherapy programs (1, 2, 3 and 4) order will depend of the group randomized. The 10 subjects will do the three-dimensional gait analysis, muscle activity during gait, evaluation of mobility, static and functional balance, and mobility tests.
  Other Names: MR4 device - device that combines super-pulsed lasers, and red and infrared LEDs (Multi Radiance Medical, Solon, OH, USA)

SUMMARY:
Hemiparesis and/or hemiplegia is one of the most common clinical signs of stroke, characterized by partial or complete loss of motor function, resulting in varying degrees of impairment and disability. The aim of this study is evaluate the acute effects of application of phototherapy to detect if this therapeutic approach may be beneficial in gait and balance post-stroke individuals. For such, 10 volunteers, with a history of injury (stroke) between 6 months to 5 years, with deficit in functional capacity in the gait due spasticity of extensor muscles of the affected limb, specifically the Triceps Sural. The evaluation will consist of three-dimensional gait analysis, muscle activity during gait, mobility, static and functional balance, and mobility of volunteers.

DETAILED DESCRIPTION:
This is a clinical, randomized, placebo-controlled, crossover and triple-blind study. Ten participants with injury history (stroke) will perform the protocol. The intervention will be held once a week for 4 weeks. Each week a different dose of phototherapy (Placebo, 10J, 30J and 50J) will be applied. The phototherapy, active or placebo, will be applied in 9 different points of anterior muscle of the thigh, 6 different points of posterior muscle of the thigh and 2 different points of the gastrocnemius muscle, bilaterally, before the tests. Only one investigator, that will not participat in any phase of the assessments sessions, will know about what program is active or placebo in phototherapy device. Randomisation will occur by a simple drawing of lots (A, B, C, or D) in the first visit. The phototherapy unit emitted the same sound regardless of the program used, active or placebo. For three-dimensional gait assessment and muscle activity will be used a SMART-D system 140® - BTS Engineering with six cameras, two Kistler force platforms Platform model 9286BA and FREEEMG® electromyography - BTS Engineering wireless system with four channels. In addition, the evaluation will quantify the static balance (force platform), the functional balance (Berg Balance Scale) and mobility (6 minute walk test and go upand team test).

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic adults with a single stroke event, with crural predominance;
* Injury (stroke) from 6 months to 5 years;
* Aged between 40 and 60 years old;
* In treatment at the Uninove physical therapy clinic;
* Able to walk barefoot, with or without support;
* With verbal comprehension, controlled systemic disease and clinically stable;
* Able to perform the 6-minute walk test.

Exclusion Criteria:

* Subjects with fixed deformities, previous surgery, previous osteoarticular dysfunction, any disease that influences the performance of the march;
* Cognitive impairment detrimental to the tests;
* Subjects who do not fit the inclusion criteria.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Three-dimensional gait assessment | The test will be performed for five weeks
  The test will collect the kinetic data of gait, records the pressure center shifts and the foot contact time with the surface of platform.

SECONDARY OUTCOMES:
Stabilometric assessment | The test will be performed for five weeks, twice a week, on the same day and time of the week.
  The test will evaluate the static balance, on the force platform.
Functional balance assessment | The test will be performed for five weeks, twice a week, on the same day and time of the week.
  The functional assessment will be composed for one test: Berg Balance Scale (BBS). The BBS is a widely used clinical test developed for evaluate of a persons static and dynamic balance abilities, for functional balance tests,is generally considered the gold standard. The scale comprises a test with a set of 14 simple balance related tasks, ranging from standing up from a sitting position, to standing on one foot. The degree of success in achieving each task is given a score of 0 (unable) to 4 (independent), and the final measure is the sum of all of the scores, it test takes 10 - 15 minutes. The interpretation of the results is: ≤20 limited data from subjects, that suggest that the tool might have similar absolute reliability at the low and high ends. Normal values = People aged 69 years without any health conditions likely to affect mobility can be expected to have a BBS score of 56/56. This normal value declines with increasing age, at a rate of 0.75 points per year.
Static and dynamic balance assessment | The test will be performed for five weeks, twice a week, on the same day and time of the week.
  The static and dynamic balance assessment will be composed for one test: Timed up and go test - test used to evaluate a person's mobility and requires static and dynamic balance.
Functional mobility assessment | The test will be performed for five weeks, twice a week, on the same day and time of the week.
  The functional mobility assessment will be composed for one test: 6-minute walk test (6MWT) - The 6MWT is used as a one-time measure of functional mobility status of patients. It's a practical test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians for the evaluation of functional exercise capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto P Leal Junior, PhD, Study Director — University of Nove de Julho
Locations (1):
- Nove de Julho University, São Paulo, Brazil

REFERENCES:
- [Background] Leal-Junior EC, Vanin AA, Miranda EF, de Carvalho Pde T, Dal Corso S, Bjordal JM. Effect of phototherapy (low-level laser therapy and light-emitting diode therapy) on exercise performance and markers of exercise recovery: a systematic review with meta-analysis. Lasers Med Sci. 2015 Feb;30(2):925-39. doi: 10.1007/s10103-013-1465-4. Epub 2013 Nov 19. PMID 24249354
- [Background] Antonialli FC, De Marchi T, Tomazoni SS, Vanin AA, dos Santos Grandinetti V, de Paiva PR, Pinto HD, Miranda EF, de Tarso Camillo de Carvalho P, Leal-Junior EC. Phototherapy in skeletal muscle performance and recovery after exercise: effect of combination of super-pulsed laser and light-emitting diodes. Lasers Med Sci. 2014 Nov;29(6):1967-76. doi: 10.1007/s10103-014-1611-7. Epub 2014 Jun 19. PMID 24942380